CLINICAL TRIAL: NCT03658044
Title: SMOP - Social Media on Prescription, a Randomised Controlled Trial
Brief Title: Social Media on Prescription for Colorectal Cancer Patients
Acronym: SMOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Högskolan Väst (Unknown)
Responsible Party: Principal Investigator, Eva Angenete, Associate professor, consultant surgeon, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SMOP
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized parallel group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participation in the internet forum (Experimental): Other: Patients will be encouraged to participate in an internet forum communicating with other patients at least once per week. Participation in the internet forum
  Interventions: Other: Participation in the internet forum
- No participation in the internet forum (Active Comparator): "Placebo" Patients will not be able to enter or read in the forum, but will be able to read general information on the webpage where the forum is placed.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Participation in the internet forum — Active participation in the forum with encouragement to participate on a weekly basis
  Arms: Participation in the internet forum
Other: Placebo — No intervention performed. Patients are offered to read the open pages on the website
  Arms: No participation in the internet forum

SUMMARY:
The overall aim with this study is to get a deeper understanding of the potential benefits with a health platform for patients diagnosed with colorectal cancer.

DETAILED DESCRIPTION:
This is a prospective randomized parallel group design. Consecutive patients will be recruited from participating hospitals and randomized to either "prescribed participation" or just receiving information about the platform but with no prescription.

All patients are also receiving standard care. After treatment all patients will receive information about the platform and the aim with the platform. A short demonstration of the platform will also be provided. The platform will contain general information on "Life after cancer treatment". It will be a forum to discuss with fellow-patients, both experienced and newly treated and it is also possible to address questions to health professionals. After the demonstration an information about the study will be given and patients will be asked to participate. If accepted a consent form will be presented and signed by the patients. All patients will be given an alias - a username, to be used at the platform which gives the patients confidentiality. However, as this is a research project they will be informed that their clinical data will be extracted from their patient charts. The alias will in a separate file be connected with their personal identification number. The patients randomized to intervention (prescribed participation) will be offered to contact a research nurse or researcher if they have any practical questions regarding the use of the platform. All patients will be asked to answer a questionnaire at baseline, 3, 6 and 12 months after surgery. Patients will be answering the questionnaires electronically on the platform or in a paper version sent by ordinary mail.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer diagnosis within 1 year
* Must be able to speak and read the Swedish language
* Must be able to use the health platform

Exclusion Criteria:

-Inability to speak and read the Swedish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Self empowerment measured by Cancer Behavior Inventory (CBI) scale | 12 months
  A 12-item measure of self-efficacy for coping with cancer that measures self empowerment and coping. Each question is answered on a 9 point Likert scale. The higher the score the more confident and self empowered

SECONDARY OUTCOMES:
Self empowerment measured by Cancer Behavior Inventory (CBI) scale | 3 months
  A 12-item measure of self-efficacy for coping with cancer that measures self empowerment and coping. Each question is answered on a 9 point Likert scale. The higher the score the more confident and self empowered
Compliance to treatment | 12 months
  How frequent is the forum used? Will be tested using newly developed questions in a questionnaire. There will be a scale from 1-5
Quality of life using a Likert scale question tested in several other studies | 12 months
  Using an assessment on a Likert scale 0-7 "How would you rate your QoL?"
Usability of a health care platform | 12 months
  Is the platform easy to use? Will be tested using newly developed questions with 4-6 answering options.
Generated Knowledge in Online Discussions | 3 years
  A qualitative analysis of the online discussions on the forum

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gellerstedt, Ph.D., Principal Investigator — Högskolan Väst; Eva Angenete, Ph.D., M.D., Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided